CLINICAL TRIAL: NCT06303921
Title: Center Without Walls for Imaging Proteinopathies With PET (CW2IP2): Phase I Pilot Study of Biodistribution, Metabolism, Excretion and Brain Uptake of 11C-M503
Brief Title: Study of Biodistribution, Metabolism, Excretion and Brain Uptake11C-M503
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 854681
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Tauopathies
Keywords: Positron Emission Tomography (PET); Brain MRI; Parkinson's disease (PD)
MeSH Terms: conditions — Tauopathies; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 11C-M503 PET (Experimental): Participants will undergo 11C-M503 PET scan, they may also have a brain MRI and Amyloid PET scan as well as neurological assessments.
  Interventions: Drug: 11C-M503 PET; Diagnostic Test: Brain MRI; Diagnostic Test: Amyloid PET; Behavioral: Neurological assessments

INTERVENTIONS:
Drug: 11C-M503 PET — 2 hour Positron Emission Tomography (PET) scan using new radiotracer 11C-M503
Diagnostic Test: Brain MRI — MRI scan of brain.
Diagnostic Test: Amyloid PET — PET scan with Florbetaben F18 or 11C-PiB
Behavioral: Neurological assessments — Neurological assessments, including a video interview.

SUMMARY:
The current protocol is to determine the biodistribution, metabolism, excretion and brain uptake of 11C-M503. The goal of this radiotracer is to quantify alpha-synuclein that is abnormally deposited in the brain of people with Parkinson's disease (PD). Investigators will compare uptake in participants with PD versus participants with multiple system atrophy (MSA) and progressive supranuclear palsy (PSP), as well as non-Parkinsonism volunteers. This multicenter project funded by an NIH U19 grant, is centered at U Pennsylvania (Penn, Grant PI: Robert Mach) in collaboration with U Pittsburgh (Pitt) (non-clinical site) Yale U, U of California at San Francisco (UCSF) and Washington University in St. Louis (WU). The University of Pennsylvania will act as the sIRB for this multi-center human subjects project and participants will be recruited from all sites.

DETAILED DESCRIPTION:
The current protocol is to determine the biodistribution, metabolism, excretion and brain uptake of 11C-M503. The goal of this radiotracer is to quantify alpha-synuclein that is abnormally deposited in the brain of people with Parkinson's disease (PD). Investigators will compare uptake in participants with PD versus participants with multiple system atrophy (MSA) and progressive supranuclear palsy (PSP), as well as non-Parkinsonism volunteers. This multicenter project funded by an NIH U19 grant, is centered at U Pennsylvania (Penn, Grant PI: Robert Mach) in collaboration with U Pittsburgh (Pitt) (non-clinical site) Yale U, U of California at San Francisco (UCSF) and Washington University in St. Louis (WU). The University of Pennsylvania will act as the sIRB for this multi-center human subjects project and participants will be recruited from all sites.

Participating clinical sites will recruit up to 20 people with PD, 20 with MSA, 10 with PSP and 20 healthy controls across sites with all participants ranging from 40-85 years old. Investigators will encourage equal participation of males and females.

This protocol will include up to 70 participants across all clinical sites (note that some of these participant scans performed at Penn may be used to calculate whole body biodistribution (BioD) and dosimetry. Investigators anticipate enrollment of up to 15-20 participants at each clinical site, who will undergo up to 120 minutes of dynamic brain PET scanning (with or without torso imaging, depending on the clinical site). A second IV or an arterial line may be placed, preferably in the arm contralateral to the side of injection, for blood metabolite analysis and/or radioactive counts at various times during the scanning session. These blood draw collections can be omitted at the discretion of the investigator. For participants at Penn that may be part of BioD analysis, urine may be collected at the end of the scan session. Participants will also undergo a research brain MRI that may be on a separate day from the PET.

PET imaging sessions will include an injection of ≤ 15 mCi (approximate range for most studies is anticipated to be 8 - 15 mCi at sites with a standard PET scanner or 3 - 15 at sites with a high sensitivity scanner) of 11C-M503. Biodistribution, metabolism, excretion and pilot brain uptake data will be collected and human dosimetry will be calculated from participants scanned at Penn who have whole body scans. PET scans will be collected to evaluate image quality and collect preliminary information on brain uptake of 11C-M503 in the disease cohorts and healthy controls. The safety of 11C-M503 will also be evaluated in all participants. Some participants (usually those with positive 11C-M503 PET scan) may also be asked to have an amyloid-beta (Aβ) PET scan to investigate specificity of 11C-M503.

ELIGIBILITY:
Inclusion Criteria:

* Patients in all cohorts will be male or female adults from 40 to 85 years of age.
* Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures or Participants who are deemed unable to provide informed consent must have a designated study partner present for consent and to accompany them to study visits
* Investigators will ask PD/MSA/PSP participants to agree to brain donation but this choice is not mandatory for participation in this study.
* Diagnosis-specific inclusion criteria: Clinical diagnoses will be determined by consensus committee for diagnostic agreement (PD, MSA, PSP or Healthy Control)

Exclusion Criteria:

* Females who are pregnant or breast feeding will be excluded, a urine pregnancy test will be performed in women of child-bearing potential prior to injection of 11C -M503, 11C-PiB or 18F-Florbetaben
* Forms of parkinsonism other than PD, PSP and MSA as defined above
* Major psychiatric disorder (e.g. schizophrenia or bipolar disorder) - major depressive disorder is allowed
* History of significant or ongoing alcohol abuse or substance abuse or dependence based on medical record review or self-reported
* Contraindications or inability to tolerate imaging, arterial line or IV placement or blood draw procedures in the opinion of an investigator or treating physician
* Contraindication to MRI, such as non-compatible implanted medical device
* Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician or investigator to be a condition that could compromise participant safety or successful participation in the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Organ Biodistribution or Dosimetry | 4 weeks
  Determine biodistribution of the radioactive investigational drug, 11C-M503 and calculate human dosimetry. A second IV or an arterial line may be placed in the arm contralateral to the side of injection for blood metabolite analysis and/or radioactive counts at various times during the scanning session. Biodistribution, metabolism, excretion and pilot brain uptake data will be collected and human dosimetry will be calculated.
PET Uptake of Tracer | 4 weeks
  Determine whether there is selective uptake of 11C-M503 in people with MSA compared to healthy volunteers, PD and PSP participants.

SECONDARY OUTCOMES:
Adverse Events | 4 weeks
  Adverse events will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Ilya M Nasrallah, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Washington University in St. Louis, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Early safety assessments including whole body dosimetry studies at Penn; coordinate patient selection criteria, centrally collect and serve all imaging and demographic data, coordinate tracer kinetic methods development and validation for human imaging, and coordinate all data to efficiently enable GO-NOGO decisions for candidate radiotracers. As a final check on diagnosis and specificity of candidate radiotracers, Investigators will request all patient participants to permit postmortem brain donation for autoradiography of relevant radiotracers on fresh frozen brain tissues. Additionally, this Core will interact with multiple ongoing studies with cohorts studying PD, MSA, PSP and FTD. Finally, a robust data sharing plan facilitates collaboration and use of support documents and imaging data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data shared as participants are enrolled and then final clinical report after study is completed.
Access Criteria: Dosimetry data. Dosimetry data for all compounds advanced to first-in-human trials will be provided on the website link for the Clinical Core. Since it is the intent of this U19 Center to provide information to the PET community on probes that have been validated in clinical research studies, these data will be provided once the CCOC has confirmed that a probe has met the validation criteria. This will include the results of dosimetry studies (organ, whole body, and EDE data) and, as requested, the organ radioactivity uptake, clearance curves and the dosimetry images in DICOM format.
  Imaging and Clinical Data. Links from the CCOC website will connect to XNAT and MARS to provide all de-identified clinical data, imaging data and related files including arterial blood sampling measurements. These data will be distributed upon request, as noted in the above policies for Data Sharing.